CLINICAL TRIAL: NCT02975284
Title: TASMA Extension Study: Long Term Efficacy and Safety of Bronchial Thermoplasty in Severe
Brief Title: Unraveling Targets of Therapy in Bronchial Thermoplasty in Severe Asthma (TASMA) Extension Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Prof J.T. Annema, Prof. Dr. J.T. Annema, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL53703.018.15
Record Dates: First submitted 2016-11-21; First posted 2016-11-29 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Severe Asthma
Keywords: bronchial thermoplasty; long term; interventional bronchoscopy
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two years after BT blood DNA/RNA will be retained
Oversight: Data Monitoring Committee: No

SUMMARY:
This study evaluates the longterm clinical outcomes, including safety and efficacy parameters after Bronchial Thermoplasty (BT) treatment over a period of 5 years. All patients included in de TASMA trial in the Netherlands will be asked to participate in the TASMA extension study.

ELIGIBILITY:
Inclusion Criteria:

* Subject participation in the TASMA study
* Ability and willingness to provide informed consent.
* Ability to comply with the study protocol

Exclusion Criteria:

* Subject participating in another clinical trial involving respiratory intervention which in the opinion of the investigator might interfere with the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who underwent BT treatment in the TASMA study (protocol No.NL45394.018.13) and were not lost to follow-up at the end of the 30 week pre-marked visit, and those willing to comply with the study protocol and routine visits for the duration of the study will be included. The expected number of patients included in the TASMA study is n=40. These are patients with severe asthma despite maximal asthma therapy.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-08; Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Severe exacerbations rate | measured yearly over 5 years
  exacerbations / subject / year measured yearly over 5 years will be compared to the health care utilization pre- and 6 months post BT-treatment.
Emergency room visit for respiratory symptoms rate | measured yearly over 5 years
  emergency room visits for respiratory symptoms/subject/year measured yearly over 5 years will be compared to the health care utilization pre- and 6 months post BT-treatment.
Hospitalization for respiratory symptoms rate | measured yearly over 5 years
  hospitalizations for respiratory symptoms/subject/year measured yearly over 5 years will be compared to the health care utilization pre- and 6 months post BT-treatment.

SECONDARY OUTCOMES:
Pre-and post bronchodilator forced expiratory volume at one second (FEV1) and related FEV1 % reversibility | measured yearly over 5 years
  measured yearly over 5 years compared to the parameters measured pre- and 6 months post-BT treatment
provocative concentration causing a 20% fall (PC20 ) methacholine test | measured yearly over 5 years
  measured yearly over 5 years compared to the parameters measured pre- and 6 months post-BT treatment
Fractional exhaled nitric oxide (FeNO) | measured yearly over 5 years
  measured yearly over 5 years compared to the parameters measured pre- and 6 months post-BT treatment
Airway-resistance (sRaw) mechanics | measured yearly over 5 years
  measured yearly over 5 years compared to the parameters measured pre- and 6 months post-BT treatment
Airway-conductance(sGaw) mechanics | measured yearly over 5 years
  measured yearly over 5 years compared to the parameters measured pre- and 6 months post-BT treatment
forced oscillation technique (FOT) | measured over 5 years
  measured yearly over 5 years compared to the parameters measured pre- and 6 months post-BT treatment
Asthma Control Questionnaire (ACQ) scores | measured yearly over 5 years
  measured yearly over 5 years compared to the parameters measured pre- and 6 months post-BT treatment
Asthma Quality of Life Questionnaire (AQLQ) scores | measured yearly over 5 years
  measured yearly over 5 years compared to the parameters measured pre- and 6 months post-BT treatment
Maintenance dose of oral steroids | measured yearly over 5 years
  measured yearly over 5 years compared to the parameters measured pre- and 6 months post-BT treatment
Maintenance dose of inhaled steroids | measured yearly over 5 years
  measured yearly over 5 years compared to the parameters measured pre- and 6 months post-BT treatment
Rescue medication use | measured yearly over 5 years
  measured yearly over 5 years compared to the parameters measured pre- and 6 months post-BT treatment
Airway smooth muscle (ASM) mass | 2 years after inclusion, 2,5 years after BT
  ASM mass as determined by percentage/absolute ASM surface area and distance of reticular basement membrane (RBM) to ASM layer in endobronchial biopsies
optical coherence tomography (OCT) determined changes | 2 years after inclusion, 2,5 years after BT
  OCT determined changes in structural airway remodelling as measured by changes in lumen area (Ai) and airway wall thickness (Aaw).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bonta, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academisch Medisch Centrum, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided